CLINICAL TRIAL: NCT00302263
Title: B181 Metobes-III: Weight Loss Maintenance of a New Bioactive Compound (Metobes-Long)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Metabolife (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: KF11-282523
Record Dates: First submitted 2006-03-13; First posted 2006-03-14 (Estimated); Last update posted 2006-03-14 (Estimated); Status verified 2005-08

CONDITIONS: Obesity
Keywords: Green tea; capsaicin; tyrosine; caffeine; energy expenditure; catecholamines
MeSH Terms: conditions — Obesity

INTERVENTIONS:
Drug: Metobes-compound

SUMMARY:
To investigate the 5-hour acute effect on energy expenditure, substrate oxidation and ad libitum food intake after intake of the Metobes-compound (green tea extract, capsaicin, tyrosine, caffeine). Furthermore, to investigate if the effect of the Metobes-compound can be inhibited by blocking the β-adrenergic receptors.

The effect of the Metobes-compound will be investigated by:

1. 5-hour energy expenditure and respiratory quotient (ventilated hood).
2. 5-h change in blood pressure and heart rate
3. 5-h change in sympathetic/parasympathetic ratio.
4. Ad libitum energy intake.
5. Self-reported postprandiel appetite sensations (VAS).

DETAILED DESCRIPTION:
Subjects 22 healthy Danish overweight to obese men (BMI between 25 and 35 kg/m2), 18 to 50 years of age. All subjects must be weight stable (within  3-kg) 2 months prior to study inclusion, non-smoking, non-athletic and have no daily use of medication.

Method

The study is designed as a 4-way crossover, randomised, placebo controlled, double-blind study. Each treatment will be separated by >1-week washout period. The treatments will consist of:

1. Bioactive Metobes compound (green tea extract, tyrosine, caffeine and capsaicin) without calcium together with 5 mg propranolol.
2. Bioactive Metobes compound (green tea extract, tyrosine, caffeine and capsaicin) without calcium together with 10 mg propranolol.
3. Bioactive Metobes compound (green tea extract, tyrosine, caffeine and capsaicin) without calcium together with a placebo tablet for propranolol (microcrystalline cellulose).
4. Placebo for the Metobes compound (microcrystalline cellulose) together with a placebo tablet for propranolol (microcrystalline cellulose).

On each test day body weight and composition will be assessed. All subjects will undergo a 5-h post dose assessment of energy expenditure by indirect calorimetry in a ventilated hood. Subjective appetite sensations, ECG and dual measures of blood pressure/heart rate will be assessed every 30 minutes. After completed respiratory measurements the subjects will be served an ad libitum lunch meal (pasta salad).

All subjects shall collect all urine excreted during the respiratory measurements. Urine samples will be analyzed for nitrogen content and content of catecholamines.

ELIGIBILITY:
Inclusion Criteria:

* 21 healthy Danish normal-weight to obese men (BMI between 20 and 35 kg/m2), 18 to 50 years of age. All subjects must be weight stable (within  3-kg) 2 months prior to study inclusion, non-smoking, non-athletic and have no daily use of medication.

Exclusion Criteria:

* They will be excluded if they do not meet the inclusion criteria and/or the blood pressure is above 165/95 mmHg and/or the ECG is abnormal.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22
Dates: Start 2005-01; Study Completion 2005-04

PRIMARY OUTCOMES:
Energy expenditure
substrate oxidation
catecholmamines
energy intake
subjective appetite sensations
sympathetic/parasympathetic ratio

CONTACTS AND LOCATIONS:
Overall Officials: Jens Kondrup, PhD, Principal Investigator — Department of Human Nutrition, The Royal Veterinary and Agricultural University, Denmark
Locations (1):
- Department of Human Nutrition, The Royal Veterinary and Agricultural University, Frederiksberg, Denmark